CLINICAL TRIAL: NCT00125528
Title: D-Cycloserine in the Management of Chronic Low Back Pain: A Double-Blind, Randomized, Placebo-Controlled Pilot Study
Brief Title: D-cycloserine in the Management of Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas J. Schnitzer (Other)
Responsible Party: Sponsor-Investigator, Thomas J. Schnitzer, professor, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A1159
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Low Back Pain; Pain
Keywords: chronic pain; low back pain; D-cycloserine
MeSH Terms: conditions — Low Back Pain; Pain; Chronic Pain | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): D-cycloserine 50mg bid/100mg bid/200 mg bid
  Interventions: Drug: D-cycloserine
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: D-cycloserine — D-cycloserine 50 mg bid; D-cycloserine 100 mg bid; D-cycloserine 200 mg bid
  Arms: 1
Drug: placebo — placebo bid
  Arms: 2

SUMMARY:
Pre-clinical studies in rats suggest that D-cycloserine (DCS) is effective in the management of chronic neuropathic pain. This pilot study will attempt to determine the effect of D-cycloserine in the treatment of chronic low back pain. Other aims of this study are to determine the safety of D-cycloserine in the treatment of chronic low back pain and to determine which pain measurement scales are best at measuring the efficacy of treatment.

DETAILED DESCRIPTION:
Human brain imaging studies indicate that the medial prefrontal cortex activity can predict more than 80% of the variance of chronic back pain intensity. Therefore, the investigators have hypothesized that modulation of brain activity at this site should result in analgesia. D-cycloserine has been shown to potentiate conditioned fear extinction. Based on this the investigators hypothesize that chronic neuropathic pain (back pain with radiculopathy) is partially mediated or potentiated by decreased ability to extinguish the pain memory, which the investigators hypothesize to be mediated through reward/aversion brain circuitry, and specifically through medial prefrontal cortex. They have tested this idea in pre-clinical studies and demonstrated that rats with neuropathic pain show analgesia over the long-term when treated with D-cycloserine. In humans with chronic back pain, the investigators hypothesize that D-cycloserine will enhance extinction of back pain which in turn should result in reduced emotional relevance of the pain, that is reduced suffering. It is quite possible that the overall intensity of the back pain will be unaffected, however, the associated suffering will be significantly attenuated.

This will be a double-blind, randomized, parallel group escalating dose study comparing D-cycloserine twice a day (bid) with placebo bid in patients with chronic low back pain. Subjects meeting inclusion criteria will continue baseline medications and be treated for 12 weeks with study drug: 50 mg bid DCS or matching placebo for the first 4 weeks, then 100mg bid DCS or matching placebo for 4 weeks and finally 200mg bid DCS or matching placebo for 4 weeks. Assessments of efficacy and safety will be undertaken every 2 weeks using standard, validated instruments to evaluate change in pain, function, quality of life and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Must have a history of low back pain for a minimum of 6 months with or without radiation of pain to leg or buttocks.
* Must be 18 years of age.
* Must have a visual analogue scale (VAS) pain score >50 mm
* Must be in generally stable health
* Must be willing to abstain from drinking alcohol during the course of the study.
* If female, must be post-menopausal for at least one year or practicing an accepted, highly effective method of contraception or abstinence and plan to continue either during the course of the study.
* Must be able and willing to read and understand instructions as well as questionnaires
* Must sign an informed consent document after complete explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits, potential risks, and are willing to participate.

Exclusion Criteria:

* Low back pain associated with any systemic signs or symptoms, e.g., fever, chills.
* Evidence of rheumatoid arthritis, ankylosing spondylitis, acute vertebral fractures, fibromyalgia, history of surgery or tumor in the back.
* Involvement in litigation regarding their back pain or have a disability claim or are receiving workman's compensation or seeking either as a result of their low back pain
* Neurologic disorder, including history of seizures
* Major psychiatric disorder during the past 6 months
* Moderate or severe depression as determined by the Beck Depression Inventory or any active suicidal ideation
* Significant other medical disease such as unstable diabetes mellitus, congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease, or malignancy
* Significant renal disease or severe renal insufficiency
* History of, or current, substance abuse/dependence including alcohol
* Significantly abnormal laboratory values
* Pregnant or lactating at any time during the course of the study
* Known sensitivity to D-cycloserine
* Currently taking any of the following medications: ethionamide, dilantin, isoniazid (INH), pyridoxine (vitamin B6)
* In the judgment of the investigator, unable or unwilling to follow the protocol and instructions
* Any change in medication for back pain in the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, M.D., Ph.D., Principal Investigator — Northwestern University; Vania Apkarian, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Result] Schnitzer TJ, Torbey S, Herrmann K, Kaushal G, Yeasted R, Vania Apkarian A. A randomized placebo-controlled pilot study of the efficacy and safety of D-cycloserine in people with chronic back pain. Mol Pain. 2016 Nov 15;12:1744806916678627. doi: 10.1177/1744806916678627. Print 2016. PMID 27852965
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5117251/pdf/10.1177_1744806916678627.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | D-cycloserine | Placebo
Started | 20 | 21
Completed | 18 | 20
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine | Placebo | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.65 (11.56) | 54.76 (10.84) | 54.71 (11.06)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 6 | 10 | 16
Numeric Rating Scale (NRS-11) [Mean (Standard Deviation); unit: units on a scale] — Numeric rating scale is an 11-point rating scale wherein participants rated their current lower back pain intensity on a scale from 0 to 10, with 0 meaning no pain and 10 being the worst pain possible. Thus, a lower score represents a better pain state at baseline.
  units on a scale | 6.47 (1.40) | 6.6 (1.50) | 6.54 (1.45)

OUTCOME MEASURES:

1. Primary Outcome: Change in Numeric Rating Scale (NRS-11)
Description: Change in NRS score after 6 weeks of treatment as compared to baseline. The numeric rating scale is an 11-point rating scale wherein participants rated their current lower back pain intensity on a scale from 0 to 10, with 0 meaning no pain and 10 being the worst pain possible. Thus, a larger negative number indicates positive change and a higher efficacy.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 18 | 20
units on a scale | -2.47 (0.50) | -1.55 (0.50)

2. Secondary Outcome: McGill Pain Questionnaire (MPQ)
Description: Change in MPQ score after 6 weeks of treatment as compared to baseline. The MPQ score uses a Pain Rating Index from 0 to 20 where 0 is evidence of no pain and 20 indicates the highest pain possible. A lower score is also indicative of a lower quality of pain. Thus, a larger negative number indicates positive change and therefore higher efficacy.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 18 | 20
units on a scale | -2.80 (0.66) | -1.00 (0.66)

ADVERSE EVENTS:
Arm/Group | D-cycloserine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 3/20 | 5/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine (N=20) | Placebo (N=21)
Headache (General disorders) | 1 (1) | 3 (3)
Lower Extremity Edema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Numbness/Tingling (Nervous system disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
It is not clear whether observed effects are due to escalating dose or duration of D-cycloserine use. A larger population and longer duration of treatment would be needed to determine this.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No